CLINICAL TRIAL: NCT02770924
Title: Clinical Outcomes After Bilateral Implantation of ZEISS AT LISA TRI AND TRI TORIC IOL
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Federal University of São Paulo (Other)
Collaborators: Instituto Paulista de Estudos e Pesquisa em Oftalmologia (Other); Eye Clinic Day Hospital, São Paulo (Other)
Responsible Party: Principal Investigator, Rubens Belfort Jr., Professor, Federal University of São Paulo
Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CAAE 49921915.1.0000.5505
Record Dates: First submitted 2016-05-04; First posted 2016-05-12 (Estimated); Last update posted 2017-09-14 (Actual); Status verified 2017-08

CONDITIONS: Cataract
Keywords: cataract; phacoemulsification; AT LISA TRI TORIC; IOL
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- AT LISA TRI TORIC (Experimental): All patients will be undergo to phacoemulsification with IOL implantation bilateral
  Interventions: Device: AT LISA TRI TORIC
- AT LISA TRI (Experimental): All patients will be undergo to phacoemulsification with IOL implantation bilateral
  Interventions: Device: AT LISA TRI

INTERVENTIONS:
Device: AT LISA TRI TORIC — phacoemulsification with IOL implantation
  Other Names: ZEISS AT LISA TRI TORIC
  Arms: AT LISA TRI TORIC
Device: AT LISA TRI — phacoemulsification with IOL implantation
  Other Names: ZEISS AT LISA TRI
  Arms: AT LISA TRI

SUMMARY:
The aim of this study is to evaluate the visual function of patients with bilateral implantation of the IOL trifocal ZEISS AT LISA TRI AND TRI TORIC by means of visual acuity tests with and without optical correction, sensitivity curve contrast, defocus curve and quality questionnaire visual function (VFQ-25).

DETAILED DESCRIPTION:
Twenty patients (40 eyes) diagnosed with cataracts and cataract surgery indication will be selected to participate in this study. The surgery will be performed by the same surgeon with 2 week interval between surgery the first and second eye. After approval of the research project by the Research Ethics Committee all patients should understand and sign the Informed Consent and Informed (IC) before surgery.

All patients will be operated by conventional phacoemulsification with implantation of intraocular lens provided by the manufacturer.

Patients will have five study visits, including the preoperative visit, operative visit four postoperative visits.

All patients will be submitted to the following routine assessments preoperatively and demographic patient information will be recorded and a detailed medical history will be obtained.

* VFQ-25 Questionnaire
* Identification of the dominant eye;
* Visual acuity
* Refraction
* Slit lamp examination
* Tonometry
* Self-keratometry;
* Corneal topography;
* Microscopy speculate
* Fundus examination.

In addition, all routine preoperative measures will be performed. lens power calculations should be performed on both eyes to ensure qualification (lens power within the diopter range (D) available) and prepare for surgery (getting the lens). The emmetropia (± 0.5 D) should be the target of patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients older than 50 years
* Cataract diagnosis indicating surgery in both eyes
* Corneal astigmatism to 12D (AT lisa tri toric)
* Corneal astigmatism less than 0,75D (AT lisa tri)
* Ability to provide consent and clarification for study participation

Exclusion Criteria:

* Significant irregular corneal astigmatism as shown by Corneal topography;
* Corneal astigmatism up 12D
* Patients diagnosed with severe visual degenerative disorders (e.g. macular degeneration or other disorder of the retina)
* Previous corneal surgery;
* Amblyopia
* Planning for multiple procedures, including IRL, LASIK, etc. during surgery or during the study
* Endothelial dystrophy clinically significant cornea (eg, Fuchs dystrophy)
* Corneal disease activity (eg, herpes simplex, herpes zoster, etc.)
* Severe diabetic retinopathy
* Retinal detachment
* Glaucoma
* Patients presenting illness or acute conditions or chronic severe that in the opinion of the investigator, would increase the surgical risk or confound the research results
* Any patient who is taking part in another study involving ocular surgery

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2016-05; Primary Completion 2017-07 (Actual); Study Completion 2017-09-13 (Actual)

PRIMARY OUTCOMES:
Binocular visual acuity for far, intermediate and near distance | Changes from Pre-Op to Month 3
  Visual acuity measurements

SECONDARY OUTCOMES:
Defocus Curve | Month 3
  Test of Defocus Curve
Contrast Sensitivity | Changes from Pre-Op and Month 3
  Compare scores of contrast sensitivity pre-op and post-op
VFQ-25 Questionnaire | Changes from Pre-Op and Month 3
  Compare answers between pre-op and post-op

CONTACTS AND LOCATIONS:
Overall Officials: Rubens Belfort, MD, PhD, Study Director — IPEPO Instituto Paulista de Estudos e Pesquisas em Oftalmologia
Locations (2):
- Brazil (2):
  - IPEPO, São Paulo
  - Eye Clinic, São Paulo

IPD SHARING:
Plan to Share IPD: Yes
paper publication